CLINICAL TRIAL: NCT06613750
Title: Comparative Efficacy and Safety of Sitagliptin Plus Gliclazide SR Versus Metformin in Treatment-Naïve Type 2 Diabetes Patients: A Randomized Non-Inferiority Study
Brief Title: Comparative Study of Sitagliptin and Gliclazide With Metformin in Type 2 Diabetes Patients With Glucotoxicity
Acronym: SG Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhibin Xu (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor-Investigator, Zhibin Xu, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFKY20240301
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus; Glucotoxicity
Keywords: Sitagliptin; Gliclazide; Metformin; Randomized Controlled Trial; Non-Inferiority Study; Glycemic Control; β-Cell Function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Gliclazide; Metformin

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized, controlled, non-inferiority study comparing the efficacy and safety of Sitagliptin Phosphate combined with Gliclazide sustained-release tablets versus Metformin in treatment-naïve patients with Type 2 Diabetes Mellitus and glucotoxicity. Participants will be randomly assigned to one of two treatment arms and followed for 12 months to evaluate glycemic control and safety outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin and Gliclazide Group (Experimental): Participants in this arm will receive sitagliptin phosphate 100 mg once daily combined with gliclazide sustained-release tablets 30-120 mg once daily for 12 weeks.
  Interventions: Drug: Sitagliptin and Gliclazide
- Metformin Group (Active Comparator): Participants in this arm will receive metformin 500 mg to 2000 mg per day, divided into two doses, for 12 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin and Gliclazide — Participants in this arm will receive sitagliptin phosphate 100 mg once daily combined with gliclazide sustained-release tablets 30-120 mg once daily for 12 weeks
  Arms: Sitagliptin and Gliclazide Group
Drug: Metformin — Participants in this arm will receive metformin 500 mg to 2000 mg per day, divided into two doses, for 12 weeks
  Arms: Metformin Group

SUMMARY:
This study compares the efficacy and safety of sitagliptin phosphate combined with gliclazide sustained-release tablets versus metformin in treatment-naïve patients with type 2 diabetes mellitus (T2DM) and glucotoxicity. The trial assesses glycemic control, patient compliance, and adverse events over a 12-week period using a randomized controlled design to determine the non-inferiority of the combined treatment.

DETAILED DESCRIPTION:
In this single-center, prospective, randomized controlled non-inferiority study, treatment-naïve patients with T2DM and glucotoxicity were enrolled to evaluate the comparative efficacy and safety of two therapeutic regimens. The study investigates the combination of sitagliptin phosphate with gliclazide sustained-release tablets against metformin alone. Participants were randomized and monitored for 12 weeks, with primary outcomes focusing on fasting plasma glucose (FPG) levels, body weight changes, and hypoglycemic events. The study also explores the impact of treatment on β-cell function and insulin sensitivity, utilizing pharmacogenomic analysis to evaluate genetic factors influencing treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM) and glucotoxicity.
* Body Mass Index (BMI) between 18 and 30 kg/m².
* Fasting plasma glucose (FPG) levels ≥ 200 mg/dL and glycated hemoglobin (HbA1c) ≥ 9.0%.
* Normal hepatic and renal functions (ALT and AST ≤ 2.5 times the upper limit of normal; serum creatinine within normal limits).
* Capable of adhering to the prescribed anti-diabetic regimen and dietary guidelines.

Exclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus.
* Hepatic or renal dysfunction (serum creatinine > 1.2 times the upper limit of normal).
* Prior use of hypoglycemic medications before screening.
* History of severe ketosis, ketoacidosis, or hyperosmolar hyperglycemic state.
* Current treatment with corticosteroids, immunosuppressive agents, or cytotoxic drugs.
* Major systemic diseases (e.g., cardiovascular, respiratory, neurological).
* Pregnant or breastfeeding women.
* Known allergies to sitagliptin or gliclazide.
* Poor compliance potential as assessed by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) Levels from Baseline to 12 Weeks | 12 weeks
  This outcome measures the change in HbA1c levels in participants over a 12-week period, comparing sitagliptin and gliclazide treatments with metformin for type 2 diabetes mellitus patients with glucotoxicity.

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) and Body Mass Index (BMI) | 12 weeks
  Secondary outcomes include changes in FPG, BMI, and the proportion of participants achieving FPG levels below 6.1 mmol/L and 7.2 mmol/L after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China